CLINICAL TRIAL: NCT00700037
Title: Effect of Atorvastatin Therapy on Fibrous Cap Thickness in Coronary Atherosclerotic Plaque as Assessed by Optical Coherence Tomography
Brief Title: Change in Plaque Characteristics With Atorvastatin
Acronym: EASY-FIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Shigeho Takarada, MD, PhD, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: wakayamamu08-001
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Acute Coronary Syndrome; Atherosclerosis; Dyslipidemia
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis; Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Atorvastatin 20mg
  Interventions: Drug: high-dose atorvastatin
- 2 (Active Comparator): atorvastatin 5mg
  Interventions: Drug: low-dose atorvastatin

INTERVENTIONS:
Drug: high-dose atorvastatin — 20mg/day
  Other Names: Lipitor20
  Arms: 1
Drug: low-dose atorvastatin — 5mg/day
  Other Names: Lipitor5
  Arms: 2

SUMMARY:
To examine effects of intensive lipid lowering therapy with atorvastatin on stabilization of coronary plaque by using optical coherence tomography (OCT) in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
Patients with acute coronary syndrome (myocardial infarction or unstable angina) who will undergo PCI and have at least one atherosclerotic lesion of >25% stenosis other than culprit lesions of current ACS are enrolled. Fibrous cap thickness of a target coronary plaque is evaluated by optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome (myocardial infarction or unstable angina) who will undergo PCI.
* plasma LDL cholesterol levels : >=100mg/dL and ≤160mg/dL
* at least one atherosclerotic lesion of >25% stenosis other than culprit lesions of current ACS

Exclusion Criteria:

* Patients who will undergo coronary bypass surgery.
* Patients with major complications during treatment of culprit coronary lesions.
* Patients with an atherosclerotic lesion with >50% stenosis at a left main trunk.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Fibrous cap thickness by OCT | 12 months

SECONDARY OUTCOMES:
macrophage number | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Akasaka, Principal Investigator — Wakayama Medical University
Locations (1):
- Wakayama Medical University, Wakayama, Wakayama, Japan

REFERENCES:
- [Derived] Komukai K, Kubo T, Kitabata H, Matsuo Y, Ozaki Y, Takarada S, Okumoto Y, Shiono Y, Orii M, Shimamura K, Ueno S, Yamano T, Tanimoto T, Ino Y, Yamaguchi T, Kumiko H, Tanaka A, Imanishi T, Akagi H, Akasaka T. Effect of atorvastatin therapy on fibrous cap thickness in coronary atherosclerotic plaque as assessed by optical coherence tomography: the EASY-FIT study. J Am Coll Cardiol. 2014 Dec 2;64(21):2207-17. doi: 10.1016/j.jacc.2014.08.045. Epub 2014 Nov 24. PMID 25456755